CLINICAL TRIAL: NCT02336698
Title: Randomized, 16-Week, Multi-Phase, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Fulranumab as Monotherapy in Subjects With Signs and Symptoms of Osteoarthritis of the Hip or Knee
Brief Title: Study of Efficacy, Safety of Fulranumab Monotherapy for OA of Hip or Knee, PAI3002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100069; 42160443PAI3002 (Other: Janssen Research & Development, LLC); 2014-003879-37 (EudraCT Number)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis; Pain
Keywords: Osteoarthritis; Pain; Fulranumab; JNJ-42160443; Monotherapy; Hip; Knee; Joint replacement surgery
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks).
  Interventions: Drug: Placebo
- Fulranumab 1 mg (Experimental): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks).
  Interventions: Drug: Fulranumab 1 mg
- Fulranumab 3 mg (Experimental): Participants will receive 4 subcutaneous (SC) injections (one injection every 4 weeks).
  Interventions: Drug: Fulranumab 3 mg

INTERVENTIONS:
Drug: Placebo — Placebo will be administered once every 4 weeks for 16 weeks by subcutaneous (SC) injection (injection under the skin) into the thigh or abdomen.
  Arms: Placebo
Drug: Fulranumab 1 mg — Fulranumab will be administered once every 4 weeks for up to 16 weeks by SC injection into the thigh or abdomen.
  Arms: Fulranumab 1 mg
Drug: Fulranumab 3 mg — Fulranumab will be administered once every 4 weeks for up to 16 weeks by SC injection into the thigh or abdomen.
  Arms: Fulranumab 3 mg

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of fulranumab as Monotherapy compared with placebo in participants with signs and symptoms of osteoarthritis of the hip or knee that are not adequately controlled by current pain therapy.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled (an inactive substance is given to one group of participants while active drug is given to another group of participants to see if there is a difference in response), parallel-group (study drugs given to participants in all treatment groups during the same time period) to evaluate the efficacy (capacity of the investigational drug to produce an effect), safety, and tolerability of fulranumab administered as monotherapy (alone; not in combination with other drug therapy) to participants with chronic moderate to severe pain and functional impairment from knee or hip osteoarthritis (OA) that is not adequately controlled by current pain therapy. The duration of participation in the study for an individual participant will be up to 67 weeks (includes a screening period of 3 weeks, a double-blind treatment period of 16 weeks, and a post-treatment follow-up period of up to 48 weeks).). All participants will be randomly assigned in a 1:1:1 ratio to 1 of 3 treatments (placebo, fulranumab 1mg, fulranumab 3mg) and given a single injection subcutaneously (under the skin) once every 4 weeks for up to 16 weeks. Blood samples will be collected from each participant at time points during the study. Safety evaluations will include assessment of adverse events, physical examinations, laboratory tests and vital signs which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis (OA) of hip or knee based on criteria defined by the American College of Rheumatology and radiographic evidence of OA (Kellgren-Lawrence class ≥2) of the study joint
* Scheduled joint replacement or planning to undergo a joint replacement surgery for the study joint
* Must have an unsatisfactory response (inadequate efficacy or poor tolerability) that includes all 3 classes of analgesic medications (acetaminophen/paracetamol, NSAID, and an opioid); For participants in the USA and Canada: Must have an unsatisfactory response (inadequate efficacy or poor tolerability) that includes all 3 classes of analgesic medications (acetaminophen/paracetamol, NSAIDs, and opioids other than codeine or codeine combination products)
* Moderate to severe pain and functional impairment based on the NRS, WOMAC pain and physical function subscales, and PGA
* During treatment and within 24 weeks after the last injection of study drug: if female of childbearing potential, is not pregnant, breast-feeding, or planning to become pregnant, or if male, will not father a child

Exclusion Criteria:

* Increased risk of osteonecrosis (ON) or rapidly progressive osteoarthritis (RPOA)
* Unstable or progressive neurologic disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of Week 16 in Western Ontario and McMaster University Arthritis Index (WOMAC) pain subscale score | Baseline, Week 16
  The WOMAC 3.1 is a multi-dimensional, osteoarthritis (OA) specific self-administered questionnaire using 24 questions with a 48-hour recall that are grouped into 3 subscales (pain, stiffness, and physical function) associated with hip or knee OA. Pain, stiffness, and physical function is rated on a scale of 0-10 (0 = less severe up to 10 = more severe).
Change from baseline to the end of Week 16 in Western Ontario and McMaster University Arthritis Index (WOMAC) physical function subscale score | Baseline, Week 16
  See WOMAC 3.1 described above.
Change from baseline to the end of Week 16 in Patient Global Assessment (PGA) score | Baseline, Week 16
  The PGA is part of a comprehensive assessment of the impact of treatment for osteoarthritis that also includes pain and physical function. The PGA included in the present study indicates the perception of osteoarthritis in the study joint at the current time. Ratings are provided on an 11-point numerical rating scale from 0 ("Very Good") to 10 ("Very Bad").

SECONDARY OUTCOMES:
Change from baseline to the end of Week 16 in Patient Global Assessment (PGA) score | Baseline, Week 16
  See PGA described above.
Change from baseline to the end of Week 16 in WOMAC Stiffness subscale score | Baseline, Week 16
  See WOMAC 3.1 described above.
Change from baseline to the end of Week 16 in daily numerical rating scale (NRS) score | Baseline, Week 16
  The numerical rating scale (NRS) uses an 11-point scale to assess OA pain ranging from 0 to 10 with high scores representing greater symptom severity (0=no pain and 10=pain as bad as you can imagine).
Change from baseline to the end of Week 16 in Medical Outcomes Study (MOS) Sleep subscale scores | Baseline, Week 16
  The MOS Sleep Scale (acute version) contains 12 items that address aspects of sleep. Six subscale scores may be calculated including: daytime somnolence, sleep disturbances, snoring, shortness of breath or headache upon awaking, adequacy of sleep and amount of sleep plus a summary index of sleep disturbances. A higher score indicates worse sleep in most domains, but the amount of sleep and adequacy of sleep are scored in the opposite direction. The primary subscale of interest in this study is daytime somnolence.
Change from baseline to the end of Week 16 in Short-Form-36 (SF-36) subscale scores | Baseline, Week 16
  The SF-36 is a self-administered, generic, 36-item questionnaire designed to cover 8 domains of functional health status and well-being, physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Scoring yields 8 subscales based on the 8 domains covered in the questionnaire. These scales are scored from 0 to 100 with higher scores indicating better health.
Change from baseline to the end of Week 16 in EuroQol, 5 dimensions, 5 levels (EQ-5D-5L) scale score | Baseline, Week 16
  The EQ-5D is a self-administered, standardized measure of health status designed to provide a generic measure of health for clinical and economic appraisal that includes the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D 5 level (5L) version will be used in this study. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and unable or extreme problems. A unique health state is defined by combining 1 level from each of the 5 dimensions.
Change from baseline to the end of Week 16 in the percentage of participants who are responders based on WOMAC pain and physical function subscale scores and PGA scale scores | Baseline, Week 16
  Responders are defined as participants with percent improvement equal to and above the threshold values for WOMAC pain and physical function subscale scores and PGA scale scores, reported separately.
Change from baseline to the end of Week 16 in the percentage of participants who are responders based on OMERACT-OARSI, MCII, and PASS scale scores | Baseline, Week 16
  Responders are defined as participants with percent improvement equal to and above the threshold values for Outcome Measures in Rheumatology initiative/Osteoarthritis Research Society International (OMERACT-OARSI), Minimal Clinically Important Improvement (MCII), and the Patient Acceptable Symptom State (PASS) scale scores.
Change from baseline to the end of Week 16 in the percentage of participants who use rescue medication and other osteoarthritis (OA) analgesia | Baseline, Week 16
  Use of rescue medication (acetaminophen/paracetamol) and other OA pain medication will be recorded weekly during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (26):
  - Phoenix, Arizona
  - Costa Mesa, California
  - Laguna Hills, California
  - Lakewood, California
  - Northridge, California
  - Santa Clarita, California
  - Thousand Oaks, California
  - Boynton Beach, Florida
  - Lake Clarke Shores, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Wichita, Kansas
  - Bay City, Michigan
  - Caro, Michigan
  - Grand Rapids, Michigan
  - Somerset, New Jersey
  - Greenville, North Carolina
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Bedford, Texas
  - Cypress, Texas
  - Houston, Texas
  - Waxahachie, Texas
  - Riverton, Utah
  - Norfolk, Virginia
- Elblag, Poland
- Spain (4):
  - A Coruña
  - Barcelona
  - Mérida
  - Santiago de Compostela
- Stourton, United Kingdom

REFERENCES:
- [Derived] Kelly KM, Sanga P, Zaki N, Wang S, Haeussler J, Louie J, Thipphawong J. Safety and efficacy of fulranumab in osteoarthritis of the hip and knee: results from four early terminated phase III randomized studies. Curr Med Res Opin. 2019 Dec;35(12):2117-2127. doi: 10.1080/03007995.2019.1653068. Epub 2019 Sep 13. PMID 31387410